CLINICAL TRIAL: NCT03299244
Title: A Multicenter, Multiple-dose, Active-controlled, Double-blind, Double-dummy Study to Compare the Therapeutic Efficacy and Safety of Oral Doses of Cinacalcet Hydrochloride With Intravenous Doses of Etelcalcetide (AMG 416) in Asian Hemodialysis Subjects With Secondary Hyperparathyroidism
Brief Title: Head-to-Head Study of Etelcalcetide and Cinacalcet in Asian Hemodialysis Patients With Secondary Hyperparathyroidism (SHPT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20150238
Record Dates: First submitted 2017-09-15; First posted 2017-10-03 (Actual); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — etelcalcetide hydrochloride; Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized by Interactive Voice Response (IVR)/Interactive Web Response (IWR) in a 1:1 ratio to either three times per week (TIW) intravenous (IV) etelcalcetide (and daily oral placebo tablets) or daily oral cinacalcet tablets (and TIW IV placebo) in a double-blind, double-dummy manner. Treatment groups will be blinded to the investigator, participants, and the Amgen study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinacalcet (Active Comparator): Participants were randomized to receive oral cinacalcet once daily and placebo intravenous (IV) bolus injection at the end of each hemodialysis session three times per week (TIW) for 26 weeks. The starting dose of cinacalcet was 25 mg daily and the dose may have been titrated at weeks 5, 9, 13, and 17 to target predialysis serum parathyroid hormone (PTH) ≤ 300 pg/mL but no lower than 100 pg/mL while maintaining corrected calcium (cCa) ≥ 8.3 mg/dL.
  Interventions: Drug: Cinacalcet
- Etelcalcetide (Experimental): Participants were randomized to receive etelcalcetide administered by intravenous bolus injection at the end of each hemodialysis session TIW and daily oral doses of placebo tablets for 26 weeks. The starting dose of etelcalcetide was 5 mg, and the dose may have been titrated at weeks 5, 9, 13, and 17 to target predialysis serum PTH ≤ 300 pg/mL but no lower than 100 pg/mL while maintaining cCa ≥ 8.3 mg/dL.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Administered intravenously three times per week.
  Other Names: AMG 416; Parsabiv®
  Arms: Etelcalcetide
Drug: Cinacalcet — Cinacalcet administered orally once a day.
  Other Names: Sensipar®; Mimpara®
  Arms: Cinacalcet

SUMMARY:
The primary objective is to demonstrate that treatment with etelcalcetide (AMG 416) is not inferior to treatment with cinacalcet for lowering serum intact parathyroid hormone (PTH) levels by > 30% from baseline among participants with chronic kidney disease (CKD) and secondary hyperparathyroidism (SHPT) who require management with hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to performing any study-related activities/procedures.
* Male or female subjects ≥ 18 years of age or older at the time of signing informed consent.
* Subject must be receiving maintenance hemodialysis 3 times weekly for at least 3 months, with adequate hemodialysis based on a delivered measure of dialysis adequacy (Kt/V) ≥ 1.2 or urea reduction ratio ≥ 65% within 4 weeks prior to screening laboratory assessments. The Kt/V formula used for a subject must be the formula used during routine care prior to screening.
* Dialysate calcium concentration must be ≥ 2.5 mEq/L (1.25 mmol/L) and stable for at least 4 weeks prior to screening laboratory assessments, and must remain ≥ 2.5 mEq/L (1.25 mmol/L) for the duration of the study.
* Subject must have SHPT as defined by one central laboratory screening predialysis serum PTH value > 500 pg/mL, within 2 weeks prior to randomization.
* Subject currently receiving vitamin D sterols must have had no more than a maximum dose change of 50% within the 4 weeks prior to screening laboratory assessments, remain stable through randomization, and be expected to maintain stable doses for the duration of the study, except for adjustments allowed per protocol or for safety reasons.
* Subject must have 1 screening predialysis serum cCa laboratory value ≥ 8.3 mg/dL measured within 2 weeks prior to randomization.
* A subject receiving calcium supplements must have had no more than a maximum dose change of 50% within 2 weeks prior to screening laboratory assessments and remain stable through randomization.
* A subject receiving phosphate binders must have had no more than a maximum dose change of 50% within the 2 weeks prior to screening laboratory assessments, remain stable through randomization, and be expected to maintain stable dose for the duration of the study, except for adjustments allowed per protocol or for safety reasons.

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study, or ≤ 30 days since ending treatment on another investigational device or drug study(s). Other investigational procedures while participating in this study are excluded.
* Subject has received etelcalcetide in a prior clinical trial of etelcalcetide.
* Subject has received cinacalcet during the 3 months prior to the first screening laboratory assessments.
* Subject has known sensitivity to any of the products or components of either cinacalcet or etelcalcetide to be administered during dosing.
* Subject has previously been randomized in this study.
* Anticipated or scheduled parathyroidectomy during the study period.
* Subject has received a parathyroidectomy within 6 months prior to dosing.
* Anticipated or scheduled kidney transplant during the study period.
* Subject has an unstable medical condition based on medical history, physical examination, and routine laboratory tests, or is otherwise unstable in the judgment of the Investigator.
* Malignancy within the last 5 years of screening (except non-melanoma skin cancers or cervical carcinoma in situ).
* Grapefruit juice is prohibited.
* Subject is pregnant or nursing, or planning to become pregnant or nurse during treatment or within 3 months after the last dose of etelcalcetide or 30 days after the last dose of cinacalcet
* Female subject of childbearing potential who is unwilling to use an acceptable method of effective contraception during treatment with investigational product (IP) through 3 months after the last dose of IP.
* Subject has a history of symptomatic ventricular dysrhythmias or Torsades de Pointes.
* Subject has a history of myocardial infarction, coronary angioplasty, or coronary arterial bypass grafting within the past 6 months prior to screening.
* Subject has clinically significant abnormalities on prestudy clinical examination or abnormalities on the most recent central laboratory tests during the screening period prior to randomization according to the Investigator including but not limited to the following:

  * serum albumin < 3.0 g/dL
  * serum magnesium < 1.5 mg/dL
  * serum transaminase (alanine transaminase [ALT] or serum glutamic pyruvic transaminase [SGPT], aspartate aminotransferase [AST] or serum glutamic oxaloacetic transaminase [SGOT]) > 3 times the upper limit of normal (ULN) at screening.
* Subject likely not available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and Investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the Investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (54):
- China (23):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Lanzhou, Gansu
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Zhanjiang, Guangdong
  - Research Site, Nanning, Guangxi
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Changzhou, Jiangsu
  - Research Site, Nanjing, Jiangsu
  - Research Site, Wuxi, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Dalian, Liaoning
  - Research Site, Shenyang, Liaoning
  - Research Site, Xi'an, Shaanxi
  - Research Site, Qingdao, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Ürümqi, Xinjiang
  - Research Site, Hangzhou, Zhejiang
- Hong Kong (3):
  - Research Site, Hong Kong
  - Research Site, Kowloon
  - Research Site, New Territories
- India (11):
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Nadiād, Gujarat
  - Research Site, Belagavi, Karnataka
  - Research Site, Mysuru, Karnataka
  - Research Site, Kozhikode, Kerala
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Chandigarh, Punjab
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Dehradun, Uttarakhand
  - Research Site, Wardha
- Malaysia (4):
  - Research Site, Ipoh, Perak
  - Research Site, George Town, Pulau Pinang
  - Research Site, Kuching, Sarawak
  - Research Site, Batu Caves, Selangor (incl. Putrajaya)
- South Korea (5):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Gumi-si, Gyeongsangbuk-do
  - Research Site, Guri-si, Gyeonggi-do
  - Research Site, Seoul
- Taiwan (8):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Keelung
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 84 centers including mainland China (43 centers), Hong Kong (2 centers), India (12 centers), South Korea (11 centers), Malaysia (4 centers), and Taiwan (12 centers). Participants were enrolled from 15 May 2018 to 12 September 2019.
Pre-assignment Details: Participants were randomized 1:1 to receive etelcalcetide or cinacalcet. Randomization was stratified by screening serum parathyroid hormone (PTH) level (< 900 pg/mL, ≥ 900 pg/mL) (< 95.40 pmol/L, ≥ 95.40 pmol/L), screening serum corrected calcium (cCa) measured by the central laboratory (≥ 9.0 mg/dL, < 9.0 mg/dL) (≥ 2.25 mmol/L, < 2.25 mmol/L), and country (China versus non-China).
Groups:
- Cinacalcet: Participants were randomized to receive oral cinacalcet once daily and placebo intravenous (IV) bolus injection at the end of each hemodialysis session three times per week (TIW) for 26 weeks. The starting dose of cinacalcet was 25 mg daily and could have been titrated at weeks 5, 9, 13, and 17 to target predialysis serum PTH ≤ 300 pg/mL but no lower than 100 pg/mL while maintaining cCa ≥ 8.3 mg/dL.
- Etelcalcetide: Participants were randomized to receive etelcalcetide administered by IV bolus injection at the end of each hemodialysis session TIW and daily oral doses of placebo tablets for 26 weeks. The starting dose of etelcalcetide was 5 mg, and could have been titrated at weeks 5, 9, 13, and 17 to target predialysis serum PTH ≤ 300 pg/mL but no lower than 100 pg/mL while maintaining cCa ≥ 8.3 mg/dL.
Period: Overall Study
Arm/Group | Cinacalcet | Etelcalcetide
Started | 317 | 320
Received Treatment | 315 | 318
Completed | 270 | 282
Not Completed | 47 | 38
Not completed — Withdrawal by Subject | 34 | 29
Not completed — Decision by Sponsor | 4 | 5
Not completed — Death | 9 | 4

BASELINE CHARACTERISTICS:
Population: The full analysis set includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cinacalcet | Etelcalcetide | Total
Number analyzed (Participants) | 317 | 320 | 637
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.9) | 52.2 (13.4) | 51.8 (13.1)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 264 | 262 | 526
  65 - 74 years | 45 | 47 | 92
  75 - 84 years | 8 | 9 | 17
  ≥ 85 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 142 | 280
  Male | 179 | 178 | 357
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian Indian | 19 | 19 | 38
  Chinese | 262 | 270 | 532
  Other | 36 | 31 | 67
Stratification Factor: Screening Intact Parathyroid Hormone (iPTH) [Count of Participants; unit: Participants]
  < 900 pg/mL | 128 | 131 | 259
  ≥ 900 pg/mL | 189 | 189 | 378
Stratification Factor: Screening Corrected Calcium (cCa) [Count of Participants; unit: Participants] — When albumin was < 4.0 g/dL (40 g/L), the calcium level was corrected according to the following formula:
  cCa (mg/dL) = total Ca (mg/dL) + (4 - albumin [g/dL]) x 0.8.
  Participants
    < 9 mg/dL | 62 | 64 | 126
    ≥ 9 mg/dL | 255 | 256 | 511
Stratification Factor: Country/Region [Count of Participants; unit: Participants]
  China | 189 | 191 | 380
  Non-China | 128 | 129 | 257
Intact Parathyroid Hormone Level [Mean (Standard Deviation); unit: pg/mL] | 1299.01 (830.99) | 1299.91 (853.82) | 1299.46 (841.87)
Corrected Calcium Level [Mean (Standard Deviation); unit: mg/dL] | 9.71 (0.75) | 9.73 (0.90) | 9.72 (0.83)
Phosphorus Level [Mean (Standard Deviation); unit: mg/dL] | 6.67 (1.61) | 6.62 (1.55) | 6.64 (1.58)
Corrected Calcium Phosphorus Product (cCa x P) [Mean (Standard Deviation); unit: mg²/dL²] | 64.70 (16.39) | 64.41 (16.33) | 64.56 (16.35)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With > 30% Reduction From Baseline in Mean Predialysis Intact Parathyroid Hormone During the Efficacy Assessment Phase - Non-inferiority Analysis
Description: Predialysis intact parathyroid hormone (iPTH) levels were measured by a central laboratory.
Time Frame: Baseline and the efficacy assessment phase (EAP; defined as weeks 20 to 27, inclusive).
Population: Full analysis set; participants with iPTH data during the EAP.
Measure: Number; unit: percentage of participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 278 | 295
percentage of participants | 66.2 | 71.9
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; The analysis was conducted on the full analysis set (637 participants). Imputation under the non-inferiority null method was applied to participants who did not have PTH data during the EAP. The Mantel-Haenszel estimator was used to calculate the treatment (Cinacalcet - Etelcalcetide), stratified by screening PTH level (< 900 pg/mL, ≥ 900 pg/mL), screening serum cCa (< 9.0 mg/dL, ≥ 9.0 mg/dL) measured by the central laboratory, and country (China versus non-China); Test type: Non-Inferiority — Etelcalcetide was considered non-inferior if the upper bound of the two-sided 95% confidence interval of the treatment difference (Cinacalcet - Etelcalcetide) was smaller than 12%, or if the lower bound of (Etelcalcetide - Cinacalcet) greater than -12%. If this criterion was met, the 2 key secondary endpoints were tested sequentially. If both key secondary endpoints were statistically significant, the other secondary endpoints were to be formally tested at an overall significance level of 0.05; Treatment Difference = 4.52, 95% CI 2-sided [-3.05 to 12.09] — Treatment difference (Etelcalcetide - Cinacalcet) stratified by screening iPTH level, screening cCa level, and country/region

2. Secondary Outcome: Percentage of Participants With > 50% Reduction From Baseline in Mean Predialysis iPTH During the Efficacy Assessment Phase
Description: Predialysis intact parathyroid hormone levels were measured by a central laboratory.
Time Frame: Baseline and the efficacy assessment phase (weeks 20 to 27, inclusive).
Population: Full analysis set; participants were considered non-responders if they did not have PTH data during the EAP (non-responder imputation).
Measure: Number; unit: percentage of participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 317 | 320
percentage of participants | 41.6 | 59.1
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; Test type: Superiority — Testing of this key secondary efficacy endpoint at an overall significance level of 0.05 was to be performed if non-inferiority was demonstrated for the primary endpoint; p < 0.001, Cochran-Mantel-Haenszel; CMH test stratified by screening iPTH level, screening cCa level, and country/region; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.47 to 2.77] — Odds ratio (Etelcalcetide : Cinacalcet) stratified by screening iPTH level, screening cCa level, and country/region

3. Secondary Outcome: Percentage of Participants With > 30% Reduction From Baseline in Mean Predialysis iPTH During the Efficacy Assessment Phase - Superiority Analysis
Description: Predialysis intact parathyroid hormone levels were measured by a central laboratory.
Time Frame: Baseline and the efficacy assessment phase (weeks 20 to 27, inclusive)
Population: Full analysis set; participants were considered non-responders if they did not have PTH data during the EAP.
Measure: Number; unit: percentage of participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 317 | 320
percentage of participants | 58.0 | 66.3
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; Test type: Superiority — Testing of this key secondary efficacy endpoint at an overall significance level of 0.05 was to be performed if non-inferiority was demonstrated for the primary endpoint, and superiority was demonstrated for the previous key secondary endpoint; p = 0.033, Cochran-Mantel-Haenszel; CMH test stratified by screening iPTH level, screening cCa level, and country/region; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.03 to 1.96] — Odds ratio (Etelcalcetide : Cinacalcet) stratified by screening iPTH level, screening cCa level, and country/region

4. Secondary Outcome: Percent Change From Baseline in Mean Predialysis Corrected Calcium During the Efficacy Assessment Phase
Description: Predialysis corrected calcium was measured by a central laboratory.
Time Frame: Baseline and the efficacy assessment phase (weeks 20 - 27, inclusive)
Population: Full analysis set; participants with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 277 | 295
percent change | -8.00 (0.50) | -10.69 (0.53)
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; Test type: Superiority; p < 0.001, Mixed-effects Model Repeated Measures; Model includes treatment group, randomization stratification factors, study week, and study week by treatment as covariates; Difference in Least Squares Means = -2.82, 95% CI 2-sided [-4.14 to -1.50], Standard Error of Mean 0.67 — Treatment difference (Etelcalcetide - Cinacalcet) stratified by screening iPTH level, screening cCa level, and country/region. Standard error of the mean is the standard error of the least squares means difference

5. Secondary Outcome: Percentage of Participants With Mean Predialysis Serum Phosphorus ≤ 4.5 mg/dL During the Efficacy Assessment Phase
Description: Predialysis serum phosphorus was measured by a central laboratory.
Time Frame: Efficacy assessment phase (weeks 20 - 27, inclusive)
Population: Full analysis set; participants with no phosphorus assessments during the EAP were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 317 | 320
percentage of participants | 26.2 | 29.1
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; Test type: Superiority; p = 0.41, Cochran-Mantel-Haenszel; CMH test stratified by screening iPTH level, screening cCa level, and country/region; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.82 to 1.65] — Odds ratio (Etelcalcetide : Cinacalcet) stratified by screening iPTH level, screening cCa level, and country/region

6. Other Pre Specified Outcome: Number of Participants With cCa < 8.3 mg/dL At Any Time During the Study
Description: Corrected calcium was measured by the central laboratory.
Time Frame: From first dose of study drug to end of study; up to 26 weeks + 30 days.
Population: Participants in the safety analysis set with at least 1 post-baseline cCa value.
  The safety analysis set includes all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 310 | 317
Participants | 245 | 273

7. Other Pre Specified Outcome: Number of Participants With cCa < 8.0 mg/dL At Any Time During the Study
Description: Corrected calcium was measured by the central laboratory.
Time Frame: From first dose of study drug to end of study; up to 26 weeks + 30 days.
Population: Participants in the safety analysis set with at least 1 post-baseline cCa value.
Measure: Count of Participants; unit: Participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 310 | 317
Participants | 194 | 241

8. Other Pre Specified Outcome: Number of Participants With cCa < 7.5 mg/dL At Any Time During the Study
Description: Corrected calcium was measured by the central laboratory.
Time Frame: From first dose of study drug to end of study; up to 26 weeks + 30 days.
Population: Participants in the safety analysis set with at least 1 post-baseline cCa value.
Measure: Count of Participants; unit: Participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 310 | 317
Participants | 61 | 109

9. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Symptomatic Hypocalcemia During the Study
Description: Common symptoms of hypocalcemia (diminished blood calcium) include paresthesias (fingertips, toes, or perioral), fatigue, muscle cramps, irritability or anxiety, tetany (eg, carpopedal spasm, laryngospasm), Chvostek's sign, seizures, and prolonged QT interval.
Time Frame: From first dose of study drug to 30 days after last dose; up to 26 weeks + 30 days.
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 315 | 318
Participants | 15 | 35

10. Other Pre Specified Outcome: Number of Participants Who Developed Antibodies to Etelcalcetide
Description: Developing antibody incidence is defined as participants who were binding antibody positive post-baseline with a negative or no result at baseline.
Time Frame: From first dose of study drug to 30 days after last dose; up to 26 weeks + 30 days.
Population: Safety analysis set participants assigned to etelcalcetide with a post-baseline antibody result.
Measure: Count of Participants; unit: Participants
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 307
Participants | 18

11. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event is defined as any untoward medical occurrence in a clinical study participant, including worsening of a pre-existing medical condition. The event does not necessarily have a causal relationship with study treatment. The investigator assessed whether each adverse event was possibly related to study drug.
  A serious adverse event is defined as an adverse event that met at least 1 of the following serious criteria:
  * fatal
  * life threatening
  * required in-patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event
Time Frame: From first dose of study drug to 30 days after last dose; up to 26 weeks + 30 days.
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 315 | 318
Participants
  Any treatment-emergent adverse event (TEAE) | 303 | 306
  Serious adverse events | 61 | 53
  TEAEs leading to discontinuation of study drug | 15 | 9
  Fatal adverse events | 9 | 4
  Treatment-related TEAEs | 243 | 250
  Treatment-related serious adverse events | 4 | 4
  Treatment-related TEAEs leading to discontinuation of study drug | 5 | 3
  Treatment-related fatal adverse events | 1 | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after last dose (up to 26 weeks + 30 days).
Description: All-cause mortality is reported for all participants randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Cinacalcet | Etelcalcetide
All-Cause Mortality (participants affected / at risk) | 9/317 | 4/320
Serious Adverse Events (participants affected / at risk) | 61/315 | 53/318
Other Adverse Events (participants affected / at risk) | 293/315 | 294/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=315) | Etelcalcetide (N=318)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 3 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 1
Cataract (Eye disorders) | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Sudden cardiac death (General disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
Complicated appendicitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infective aneurysm (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 4 | 7
Pyelonephritis acute (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 3 | 5
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 2
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 | 1
Transplant evaluation (Investigations) | 0 | 1
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Jugular vein occlusion (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 2 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Uraemic encephalopathy (Nervous system disorders) | 1 | 0
Device malfunction (Product Issues) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 2
End stage renal disease (Renal and urinary disorders) | 2 | 3
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 1 | 0
Jejunostomy (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Granulomatosis with polyangiitis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 4
Hypotension (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Subclavian vein stenosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=315) | Etelcalcetide (N=318)
Abdominal discomfort (Gastrointestinal disorders) | 17 | 15
Constipation (Gastrointestinal disorders) | 12 | 18
Diarrhoea (Gastrointestinal disorders) | 14 | 19
Nausea (Gastrointestinal disorders) | 45 | 35
Vomiting (Gastrointestinal disorders) | 47 | 30
Chest discomfort (General disorders) | 16 | 15
Nasopharyngitis (Infections and infestations) | 31 | 28
Upper respiratory tract infection (Infections and infestations) | 33 | 34
Blood calcium decreased (Investigations) | 218 | 252
Blood calcium increased (Investigations) | 16 | 16
Blood pressure increased (Investigations) | 18 | 12
Decreased appetite (Metabolism and nutrition disorders) | 18 | 10
Hypercalcaemia (Metabolism and nutrition disorders) | 17 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 13 | 19
Hyperphosphataemia (Metabolism and nutrition disorders) | 34 | 26
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 35
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 37 | 48
Dizziness (Nervous system disorders) | 24 | 28
Hypoaesthesia (Nervous system disorders) | 8 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 16
Dialysis hypotension (Vascular disorders) | 11 | 18
Hypertension (Vascular disorders) | 18 | 16
Hypotension (Vascular disorders) | 27 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT03299244/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT03299244/SAP_001.pdf